CLINICAL TRIAL: NCT03841097
Title: A Phase IV, Prospective, Randomized, Open-label, Comparative Analysis, Single-center Study of Pulse Wave Velocity Evaluation, Tacrolimus TTR and Co-efficient of Tacrolimus Variation of African American Kidney Recipients Receiving Standard of Care Immediate Release Tacrolimus Capsules or Extended Release Tacrolimus Tablets
Brief Title: Pulse Wave Velocity, Tacrolimus Time in Therapeutic Range and CV in African American Kidney Transplants
Acronym: PTAAK
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Roy D. Bloom, MD (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Roy D. Bloom, MD, Principal Investigator, Professor of Medicine, and Medical Director of the Penn Kidney Transplant Program, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 832046
Record Dates: First submitted 2018-12-10; First posted 2019-02-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Kidney Transplant; Complications
Keywords: Renal; Transplant; Pulse wave velocity
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended Release Tacrolimus Tablets (Active Comparator): Dosed once daily in the morning and started at a dose of 0.14 mg/kg/day by the first day after kidney transplant (post-operative day 1). This medication will be given with rabbit antithymocyte globulin (rATG) induction, oral mycophenolate mofetil (MMF) and oral steroids to help prevent rejection. These medications will be ordered per standard of care both inpatient and outpatient.
  Interventions: Drug: Extended Release Tacrolimus Tablets
- Immediate Release Tacrolimus Capsules (Active Comparator): Dosed twice daily 12 hours apart and started at a dose of 0.1mg/kg/day by the first day after kidney transplant (post-operative day 1). This medication will be given with rabbit antithymocyte globulin (rATG) induction, oral mycophenolate mofetil (MMF) and oral steroids to help prevent rejection. These medications will be ordered per standard of care both inpatient and outpatient.
  Interventions: Drug: Immediate Release Tacrolimus Capsule

INTERVENTIONS:
Drug: Extended Release Tacrolimus Tablets — The primary objective is to assess the change in pulse wave velocity (PWV) and vascular compliance measurements from baseline to 12-24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
  Other Names: LCPT; Envarsus XR®
  Arms: Extended Release Tacrolimus Tablets
Drug: Immediate Release Tacrolimus Capsule — The primary objective is to assess the change in pulse wave velocity (PWV) and vascular compliance measurements from baseline to 12-24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
  Other Names: IR-TAC; Prograf®
  Arms: Immediate Release Tacrolimus Capsules

SUMMARY:
The primary purpose of this study is to evaluate the pulse wave velocity and vascular compliance measurements at the beginning and the end of the study while the participants are taking either extended release tacrolimus tablets (known by brand name Envarsus XR®, and also referred to as LCPT in this study) given once-daily each morning after transplantation or immediate release tacrolimus capsules (also known by brand name Prograf® or abbreviation IR-TAC in this study) that are administered twice-daily 12 hours apart after kidney transplantation. Pulse wave velocity and vascular compliance measurements are two non-invasive tests that are used to evaluate how well the blood vessels adapt to each heartbeat. The secondary purpose is to look at the effectiveness and safety of LCPT given once-daily compared to IR-TAC given twice-daily 12 hours apart after kidney transplantation.

DETAILED DESCRIPTION:
There are several medicines that are given to kidney transplant patients to prevent the body's immune system from rejecting (not accepting) the transplanted kidney. Frequently, more than one medicine is used at the same time to prevent rejection after kidney transplant. Some of the medicines currently used are IR-TAC, Mycophenolate mofetil (MMF), Mycophenolate sodium (MPS), and corticosteroids. IR-TAC is currently approved by the Food and Drug Administration (FDA) under the trade name of Prograf® or equivalent generic versions to prevent rejection in kidney transplant recipients. IR-TAC is taken twice daily (12 hours apart), and the dose is adjusted by the transplant provider to keep the level of tacrolimus in the blood from being too low or too high.

LCPT is a tablet containing the same active ingredient that is in IR-TAC but LCPT has been designed to release tacrolimus over a longer period of time so that it only has to be taken once a day in the morning. The dose of it is also adjusted by the transplant provider to keep the level of tacrolimus in the blood from being too low or too high. It has been approved by the FDA for prevention of rejection in kidney transplant recipients in combination with other medications to prevent rejection after kidney transplant.

In this study, the participants will be randomly assigned by chance (like flipping a coin) to receive either IR-TAC or LCPT from the time of transplant-on. Approximately half (30) of the study participants will be given IR-TAC and half will be given LCPT. Both the study participants and the transplant providers will know which medication that the participants are receiving. The participants will remain in the study for up to 12 months during which time they will be seen for monthly clinic visits, and complete labs per the standard of care.

Additionally, the study investigators will take an additional blood sample to further find out how the body absorbs and breaks down the medication tacrolimus. Participants will also undergo non-invasive pulse wave velocity and vascular compliance measurements within 3 days of post transplant, then 1 month and 12 months after transplant. Pulse wave velocity and vascular compliance measurements are two non-invasive tests that are used to evaluate how well the blood vessels adapt to each heartbeat. All participants will also be taking either Mycophenolate mofetil (MMF) or Mycophenolate sodium (MPS) and corticosteroids to prevent rejection. These procedures will help the investigators to look at the effectiveness and safety of LCPT compared to IR-TAC after kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who self-report their race/ethnicity as Black-non-Hispanic only (which may include self-reported African ancestry as African-American, Afro-Caribbean or African)
* Subjects receiving a first or second deceased donor or living donor kidney transplant at the Hospital of the University of Pennsylvania
* Subjects whose body mass index (BMI) ≥19
* Subjects who are sero-positive for Hepatitis B or C positive may also be enrolled.
* Subjects whose concurrent immunosuppression at the time of transplant will be (generic or brand formulation) Mycophenolate mofetil (MMF, CellCept) or mycophenolic sodium (MPS, Myfortic®), either a standard prenisone taper or an early withdrawal protocol, and induction with rabbit-antithymocyte globulin (Thymoglobulin®).

Exclusion Criteria:

* Subjects who are greater than 75 years old
* Known hypersensitivity to Tacrolimus and hydrogenated castor oil
* Subjects who are not self-described as being of Black African descent and living in the United States
* Subjects who self-report their race/ethnicity as Black-Hispanic or Multiracial
* Subjects who are recipients of organ transplants other than kidney
* Subjects who are recipients of third time or more kidney transplants
* Subjects who are HIV positive at the time of pre-transplant screening
* Subjects with recurrent focal segmental glomerulosclerosis (FSGS)
* Subjects with any severe medical condition (including infection or severe liver disease) requiring acute or chronic treatment that in the investigator's opinion would interfere with study participation
* Subjects with WBC ≤ 2000/mm3 or ANC ≤ 1500 mm3 with PLT ≤ 75,000/mm3 or HGB < 8 g/dL
* Subjects with mental or physical conditions or known non-adherence (defined as documentation in the patient chart of multiple missed visits and/or medication doses) which in the investigator's opinion would interfere with the objectives of the study
* Subjects who have been exposed to investigational therapy within 30 days prior to enrollment or five half-lives of the investigational product (whichever is greater).
* Subjects with severe diabetic gastroparesis or other severe GI disturbances that could interfere with Tacrolimus absorption
* Subjects who have underwent gastric bypass at any time pre transplant.
* Pregnant or nursing (lactating) women subjects, where pregnancy is defined as a state of female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml).
* Women subjects of child-bearing potential, defined as all women physiologically capable of becoming pregnant who are unwilling to use a double-barrier method of contraception, UNLESS they are
* Women whose career, lifestyle, or sexual orientation preclude intercourse with a male partner
* Women whose partners have been sterilized by vasectomy or other means

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Assess Change in Pulse Wave Velocity | baseline and months 12-24 post transplant
  To assess the change in PWV measurements (m/sec) from baseline to 12-24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Assess Change in Vascular Compliance measurements | baseline and months 12-24 post transplant
  To assess the change in vascular compliance using central blood pressure (mmHg) from baseline to 12-24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Assess Change in Vascular Compliance | baseline and months 12-24 post transplant
  To assess the change in vascular compliance using Augmentation Index (ratio) from baseline to 12 -24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.

SECONDARY OUTCOMES:
Assess Change in Pulse Wave Velocity measurements | baseline and 1 month post transplant
  To assess the change in PWV measurements (m/sec) from baseline to 1 month after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Assess Change in Vascular Compliance measurements | baseline and 1 month post transplant
  To assess the change in vascular compliance using central blood pressure (mmHg) from baseline to 1 month after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
  Augmentation Index (ratio) measurements from baseline to 1 month after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Assess Change in Vascular Compliance | baseline and 1 month post transplant
  To assess the change in vascular compliance using Augmentation Index (ratio) from baseline to 1 month after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
  Augmentation Index (ratio) measurements from baseline to 1 month after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare Percent of Kidney Recipients with Tacrolimus Time in Therapeutic Range | 1 year
  To compare % of kidney recipient subjects with Tacrolimus time in therapeutic range (TTR) < 60% or < 75% by 12-24 months: (TTR will be defined as trough level between 7.5-12.5 ug/L between week 1 after transplant-month 1, 7.5-10.5ug/L between Months 2-3, 5.5-8.5 ug/L between months 4-12 after transplant, and 4.5-7.5ug/L 12 month onward) in patients on LCPT compared to those on IR-Tac.
Compare the variability of Tacrolimus levels between LCPT and IR-Tac | First 12-24 months
  To compare the variability of Tacrolimus levels between LCPT and IR-Tac using coefficient of variation (CV); high Tacrolimus CV will be defined > 40% during the first 12-24 months after transplant in kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare steady-state mg/kg Tacrolimus dosing requirements | At baseline
  To compare steady-state mg/kg Tacrolimus dosing requirements to reach initial therapeutic troughs (defined as 8-12 ug/L) in kidney recipient subjects on LCPT compared to those on IR-Tac by CYP3A5*1 expressers vs. CYP3A5*1 non-expressers.
Compare Tacrolimus-related medication adherence | at months 1,2,3,6 and 12-24
  To compare Tacrolimus-related medication adherence (measured by patient report of missed doses at transplant nephrology visits) in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare mean systolic and arterial blood pressure | at baseline and 12-24 months post-transplant
  To compare mean systolic and arterial blood pressure in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare anti-hypertensive medication use | at baseline and 12-24 months post-transplant
  To compare anti-hypertensive medication use in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare mean diastolic and arterial blood pressure | at baseline and 12-24 months post-transplant
  To compare mean diastolic and arterial blood pressure in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare estimated glomerular filtration rate (eGFR) measured by the Modification of Diet in Renal Disease (MDRD) formula | At 6 months and 12-24 months post- transplant
  To compare estimated glomerular filtration rate (eGFR) via Modification of Diet in Renal Disease (MDRD) 4 calculation in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare hemoglobin A1C values | Post- transplant at months 3, 6, and 12-24
  To compare the occurrence of a new diagnosis pre-diabetes (as documented in the electronic health record) and hemoglobin A1C values in all non-diabetic kidney transplant subjects on LCPT compared to those on IR-Tac.
Compare the incidence of development of donor specific antibodies | At months 1, 3, 6 and 12-24 post- transplant
  To compare the incidence of development of donor specific antibodies (DSA) in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare the incidence of development of BK virus | At months 1, 3, 6, and 12-24 post- transplant
  To compare the incidence of development of BK virus (defined as BKV > 2.5 log copies/mL) in all kidney recipient subjects on LCPT compared to those on IR-Tac.
Compare the incidence of serious adverse events | At months 6 and 12-24 post- transplant
  To compare the incidence of serious adverse events (SAEs) (including infections resulting in hospitalization, development of biopsy proven cellular and antibody mediated rejection by Banff criteria when biopsy performed for clinical indications, graft loss and patient death) in all kidney recipient subjects on LCPT compared to those on IR-Tac.

CONTACTS AND LOCATIONS:
Overall Officials: Roy D Bloom, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States